CLINICAL TRIAL: NCT06072118
Title: A Multicenter, Single-arm, Clinical Trial of Adrenomedullin for Cerebral Autosomal Dominant Arteriopathy With Subcortical Infarcts and Leukoencephalopathy
Brief Title: Adrenomedullin for CADASIL
Acronym: AMCAD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cerebral and Cardiovascular Center, Japan (Other)
Responsible Party: Principal Investigator, Masafumi Ihara, Director of Neurology, National Cerebral and Cardiovascular Center, National Cerebral and Cardiovascular Center, Japan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCVC-AM-CAD; jRCT2051210117 (Registry Identifier: Japan Registry of Clinical Trials)
Record Dates: First submitted 2023-10-02; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Cadasil
MeSH Terms: conditions — CADASIL | interventions — Adrenomedullin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adrenomedullin group (Experimental)
  Interventions: Drug: Adrenomedullin

INTERVENTIONS:
Drug: Adrenomedullin — Dosing at 15 ng/kg/min for 8 hours is continued for 14 days.

SUMMARY:
Cerebral autosomal dominant arteriopathy with subcortical infarcts and leukoencephalopathy (CADASIL) is the most common form of hereditary cerebral small vessel disease, with no proven disease-modifying treatments. Adrenomedullin, a vasoactive peptide, has angiogenic, vasodilation, anti-inflammatory, and anti-oxidative properties and could have triple sites of action on components of the neuro-glial-vascular unit consisting of vessels, microglia and oligodendrocytes or, more specifically, on the white matter oligovascular unit. The aim of the AMCAD trial is to assess the safety and efficacy of Adrenomedullin in CADASIL patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have given written informed consent from the patient or the sponsor to participate in the clinical trial
2. Patients aged between 20 and 90 at the time of obtaining consent
3. Patients diagnosed as CADASIL after confirming NOTCH3 gene mutation by genetic testing
4. Patients with Mini-mental state examination-J score of 10-27 or Trail maiking test score (age ajustment) of average + 1.5 SD (standard deviation) or higher

Exclusion Criteria:

1. Patients who cannot perform cognitive function tests (deafness, blindness, etc., MMSE-J less than 10 points Severe cognitive impairment, etc.)
2. Patients received reatment with prohibited drugs or prohibited therapy within the past 12 weeks from the time of registration
3. Patients who started to take concomitant restriction drugs or changed dosage of concomitant restriction drugs within the past 4 weeks from the time of registration
4. Patients whose Mini-mental state examination-J with 4 or more points improvements between the time of registration and 4 weeks or more at the time of screening (If patients who take concomitant restriction drugs)
5. Patients with active infections requiring antibiotic treatment at registration
6. Patients with a disability equivalent to modified Rankin Scale 5 at registration
7. Patients with severe consciousness impairment (Japan Coma Scale 100 or more)
8. Patients with severe renal impairment (estimated GFR less than 30 mL / min / 1.73m2) at registration
9. Patients with severe liver damage (transaminase AST (GOT) or ALT (GPT) 100 IU / L or more) at registration
10. Patients diagnosed as having cerebral infarction or intracranial hemorrhage or transient ischemic attack or cerebral aneurysm with high probability of rupture within the last 12 weeks from the time of registration
11. Patients with occlusion or severe stenosis of the intracranial main artery or carotid artery at the time of registration
12. Patients with significant ECG abnormalities (atrioventricular block of 2-3 degrees, extension of QRS interval of 120 ms or more, extension of QTcB of 450 msec or more) at registration, or past histroy of acute coronary syndrome or acute heart failure within the last 12 weeks from the time of registration
13. Patients with systolic blood pressure less than 100 mmHg at registration
14. Patients whose pulse rate is less than 45 beats / minute or 120 beats / minute or more at registration
15. Patients with substance abuse or alcoholism
16. Patients who cannot perform MRI
17. Patients with active solid malignant tumors
18. Patients who do not give consent to contraception from the date of obtaining consent until the end of the safety evaluation period
19. Pregnant, lactating, and possibly pregnant
20. Patient who participated in another trial within 24 weeks before registration
21. Other patients judged by the Investigator or Investigator to be ineligible for this study

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2023-01-23 (Actual); Study Completion 2023-06-12 (Actual)

PRIMARY OUTCOMES:
Cerebral blood flow change rate evaluated by arterial spin labeling | at 28 days post adrenomedullin administration
  Frontal lobe

SECONDARY OUTCOMES:
Cerebral blood flow change rate evaluated by arterial spin labeling | at 8 hours / 15 days / 90 days / 180 days post adrenomedullin administration
  Frontal lobe
Cerebral blood flow change rate evaluated by arterial spin labeling | at 8 hours / 15 days / 28 days / 90 days / 180 days post adrenomedullin administration
  Whole brain mean and each area
Mean diffusivity change rate of the white matter evaluated by MR diffusion tensor imaging | at 8 hours / 15 days / 28 days / 90 days / 180 days post adrenomedullin administration
  Whole brain mean and each area
Fractional anisotropy change rate of the white matter evaluated by MR diffusion tensor imaging | at 8 hours / 15 days / 28 days / 90 days / 180 days post adrenomedullin administration
  Whole brain mean and each area
Change in times of Trail making test-A/B from baseline evaluation | at 15 days / 28 days / 90 days / 180 days post adrenomedullin administration
Change in scores of Montreal cognitive assessment from baseline evaluation | at 15 days / 28 days / 90 days / 180 days post adrenomedullin administration
Change in scores of Wechsler Adult Intelligence Scale-Fourth edition from baseline evaluation | at 15 days / 28 days / 90 days / 180 days post adrenomedullin administration
Occurence of cerebral infarction | at 8 hours / 15 days / 28 days / 90 days / 180 days post adrenomedullin administration
Cerebral blood flow change rate evaluated by single photon emission computed tomography | at 28 days post adrenomedullin administration
  Frontal lobe
Safety: Serious adverse event | From the initiation of adrenomedullin administration to 28 days post

CONTACTS AND LOCATIONS:
Locations (1):
- National Cerebral and Cardiovascular Center, Suita, Osaka, Japan

REFERENCES:
- See also: Trial registration — https://jrct.niph.go.jp/en-latest-detail/jRCT2051210117